CLINICAL TRIAL: NCT03316261
Title: Freder1k-Study - Identification of Infants With Increased Type 1 Diabetes Risk for Enrollment Into Primary Prevention Trials
Brief Title: Freder1k-Study - Testing Infants for Type 1 Diabetes Risk
Status: Recruiting | Type: Observational
Sponsor: Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Anette-Gabriele Ziegler, Director - Institute of Diabetes Research, Helmholtz Zentrum München
Other Study IDs: GPPAD-02
Record Dates: First submitted 2017-10-12; First posted 2017-10-20 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Identification of Infants at Risk for Type 1 Diabetes
Keywords: infants; type 1 diabetes; Freder1k
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Freder1k-Study will identify infants who have a high genetic risk of type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes is a common chronic disease in childhood and is increasing in incidence. Type 1 diabetes is diagnosed by hyperglycemia often in combination with symptoms of weight loss, thirst, fatigue and frequent urination, sometimes with ketoacidosis. The clinical onset is preceded by an asymptomatic phase identified by serum multiple beta-cell autoantibodies. Neonates and infants who are at increased risk to develop multiple beta-cell autoantibodies and type 1 diabetes can now be identified using genetic markers. This provides opportunity for introducing early therapies to prevent beta-cell autoimmunity and type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age: up to age 6 weeks
* provided written informed consent by custodial parent

Exclusion Criteria:

-

Ages: 1 Day to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Freder1k-Study will identify infants who have a high genetic risk of type 1 diabetes.
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
greater than 10% risk for multiple beta-cell autoantibodies/type 1 diabetes | one-time testing before age 6 weeks
  increased risk will be identified by risk scores derived from SNPs

CONTACTS AND LOCATIONS:
Overall Officials: Anette-Gabriele Ziegler, Study Chair — Helmholtz Zentrum München, IDF-1
Locations (1):
- Institut für Diabetesforschung, Helmholtz Zentrum München, Munich, Germany

REFERENCES:
- [Derived] Hippich M, Holthaus L, Assfalg R, Zapardiel-Gonzalo J, Kapfelsperger H, Heigermoser M, Haupt F, Ewald DA, Welzhofer TC, Marcus BA, Heck S, Koelln A, Stock J, Voss F, Secchi M, Piemonti L, de la Rosa K, Protzer U, Boehmer M, Achenbach P, Lampasona V, Bonifacio E, Ziegler AG. A Public Health Antibody Screening Indicates a 6-Fold Higher SARS-CoV-2 Exposure Rate than Reported Cases in Children. Med. 2021 Feb 12;2(2):149-163.e4. doi: 10.1016/j.medj.2020.10.003. Epub 2020 Oct 29. PMID 33163984
- See also: GPPAD — http://www.gppad.org